CLINICAL TRIAL: NCT02849964
Title: Factors Related to Geographical Variation in the Incidence of End-stage Renal Failure: An Analysis in 5 French Regions
Acronym: VIgIE
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Collaborators: Agence de La Biomédecine (Other Government); Central Hospital, Nancy, France (Other); University Hospital, Strasbourg, France (Other); Observatoire Régional de la Santé d'Alsace (Unknown)
Responsible Party: Sponsor
Other Study IDs: VIgIE
Record Dates: First submitted 2016-07-27; First posted 2016-07-29 (Estimated); Last update posted 2016-07-29 (Estimated); Status verified 2016-07

CONDITIONS: Renal Insufficiency
Keywords: Incidence; Renal Replacement Therapy; Socioeconomic Factors; Clinical Practice Pattern
MeSH Terms: conditions — Renal Insufficiency

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- First time renal replacement therapy: Patients beginning renal replacement therapy by renal dialysis or preemptive kidney transplant.

SUMMARY:
The REIN registry highlights significant disparities in the incidence of end-stage renal disease (ESRD) between regions, especially in the North East of France. According to the literature, the incidence of ESRD in an area could be related to contextual factors influencing the needs for dialysis or transplantation (age structure, prevalence of risk factors, socioeconomic and morbidity levels), as well as to primary and secondary care provision (general practitioners and nephrologists) and to practice patterns in nephrology.

The aims of this project are the following:

1. to compare the incidence of renal replacement therapy (dialysis or preemptive transplantation) for ESRD between the "départements" and the "cantons" belonging to the 5 regions of Eastern France (Alsace, Lorraine, Champagne-Ardenne, Bourgogne and Franche-Comté), while taking into account differences in population sizes and spatial patterns of the data,
2. to analyse the relations between incidence disparities and socioeconomic environment, geographic accessibility to primary and secondary care and medical practice patterns, after adjusting for morbidity and mortality rates (incidence of diabetes, cardiovascular mortality).

This project will enable a better understanding of the mechanisms involved in the spatial variations of ESRD incidence, while disentangling effects related to the need from effects related to service supply in different socio-economic contexts. It will be possible to identify a lack of equity in access to renal replacement therapy if, after adjusting for need indicators, there were variations of incidence of ESRD related to availability of service or to socioeconomic context. Highlighting such effects would lead to search for corrective measures in collaboration with the different stakeholders.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and older
* Resident of the 5 French administrative regions (Alsace, Bourgogne, Champagne-Ardenne, Franche-Comté, and Lorraine)
* First renal replacement therapy by renal dialysis or preemptive kidney transplant between January 1st, 2010 and December 31, 2014
* Found in the REIN registry

Exclusion Criteria:

* Transfer from another French administrative region
* Return to renal dialysis after graft rejection or a period without dialysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All person entering renal replacement therapy, either by renal dialysis or preemptive kidney transplant, between January 1st, 2010 and December 31, 2014, and residing in the study zone (5 northeastern administrative regions of France), found in the French REIN registry.
Sampling Method: Non-Probability Sample
Enrollment: 6835 (Actual)
Dates: Start 2015-09; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Factors associated with renal replacement therapy | Study period: 2010-2014
  Analysis of the association between renal replacement therapy incidence disparities and socioeconomic environment, geographic accessibility to primary and secondary care and medical practice patterns.

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth Monnet, MD, PhD, Principal Investigator — Centre d'Investigation Clinique, CHU Besançon; Carole Ayav, MD, Principal Investigator — Centre d'Investigation Clinique, CHU Nancy
Locations (4):
- France (4):
  - Centre d'Investigation Clinique, CHU de Besançon, Besançon
  - Hôpital William Morey, Néphrologie, Chalon-sur-Saône
  - CHU de Reims, Néphrologie, Reims
  - Centre d'Investigation Clinique CHU de Nancy, Vandœuvre-lès-Nancy

IPD SHARING:
Plan to Share IPD: No